CLINICAL TRIAL: NCT05306262
Title: Effects of Catalepsy on the Parasympathetic Tone Assessed by ANI (Analgesia/Nociception Index) and on Absorption, Dissociation and Perception of Time During the Hypnotic Trance.
Brief Title: Interest of Catalepsy in the Hypnotic Trance
Acronym: CATALHYPNOANI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020/03
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Hypnosis
Keywords: Hypnosis; Catalepsy; Parasympathetic tone; Absorption; Dissociation; Perception of time
MeSH Terms: conditions — Catalepsy; Dissociative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypnotic trance (Active Comparator): Hypnosis session of comfort for 20 minutes
  Interventions: Procedure: Hypnosis session
- hypnotic trance + catalepsy (Experimental): Catalepsy + Hypnosis session of comfort for 20 minutes
  Interventions: Procedure: Hypnosis session; Other: Catalepsy

INTERVENTIONS:
Procedure: Hypnosis session — Comfort hypnosis: accompaniment of a pleasant memory.
Other: Catalepsy — Catalepsy of the hand.
  Arms: hypnotic trance + catalepsy

SUMMARY:
Catalepsy seems to facilitate hypnotic induction and deepen hypnotic trance, although no work confirms the usefulness of this technique which is in common use in hypnosis. Furthermore, it has been shown that the hypnotic trance state is accompanied by an increase in parasympathetic tone, the non-invasive measurement of which is easy by the ANI monitor (Analgesia Nociception Index).

The research hypothesis is that, by adding a body dissociation, catalepsy could facilitate and intensify the hypnotic trance, the intensity of which can be monitored and is proportional to the parasympathetic tone.

DETAILED DESCRIPTION:
After randomization, subjects will either benefit from the normal hypnotic trance, or from the hypnotic trance associated with catalepsy of the hand.

T0 = installation in a sitting position and collection of an accompanying theme T1 = induction of the hypnotic trance (closing eyes) with restitution of the theme to the patient and suggestion of comfort over a period of 5 to 10 min T2 = validation of comfort by a pre-established signal T3 = return to consciousness (opening eyes) T4 = end of questionnaire about absorption, dissociation and time perception

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* Consent for participation
* Affiliation to the social security system

Exclusion Criteria:

* Arrhythmia (atrial fibrillation, pacemaker, defibrillator)
* Autonomic nervous system disorder (paraplegia, epilepsy, etc.)
* Pregnant or breastfeeding woman
* Patients under protection of the adults (guardianship, curators or safeguard of justice)
* Communication difficulties

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
Parasympathetic tone | 30 minutes
  Analgesia Nociception Index (ANI)

SECONDARY OUTCOMES:
Absorption | 30 minutes
  Numeric scale from 0 to 10 (0=not at all, 10=completely)
Dissociation | 30 minutes
  Numeric scale from 0 to 10 (0=completely in the reality, 10=completely disconnected from reality)
Time perception (minute) | 30 minutes
  Difference between the time of hypnosis session estimated by the patient and the actual time of hypnosis session (from closing to opening the eyes).
Variation of Heart Rate (beat per minute) | 30 minutes
  Heart rate measured by a pulse oximeter
Variation of Respiratory Rate (breath per minute) | 30 minutes
  Respiratory rate assessed by the investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Emergences, Rennes, France